CLINICAL TRIAL: NCT06601803
Title: Effect of Surgiphor (sterile Povidone-Iodine) Wound Irrigation on Rate of Positive Deep Culture and NGS in Primary Total Shoulder Arthroplasty- a Prospective, Randomized Pilot Study
Brief Title: Surgiphor Us in TSA
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SNAM20D1057
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Total Shoulder Arthroplasty; Shoulder Infection; Povidone Iodine
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Total Shoulder Arthroplasty washed with Saline (Active Comparator): This arm will consist of sterile normal saline to be used before and after placement of shoulder arthroplasty components
  Interventions: Drug: sterile saline solution; Procedure: Sample Collection
- Total Shoulder Arthroplasty washed with Surgiphor (Povidone Iodine) (Active Comparator): This arm will consist of Surgiphor to be used before and after placement of shoulder arthroplasty components
  Interventions: Drug: Surgiphor; Procedure: Sample Collection

INTERVENTIONS:
Drug: sterile saline solution — The shoulder will be washed with normal sterile saline before and after placing the shoulder implant
  Arms: Total Shoulder Arthroplasty washed with Saline
Drug: Surgiphor — The shoulder will be washed with Surgiphor (Povidone Iodine) before and after placing the shoulder implant
  Arms: Total Shoulder Arthroplasty washed with Surgiphor (Povidone Iodine)
Procedure: Sample Collection — During the surgical procedure, 4 swabs of the surgical wound will be taken at various times throughout the procedure

SUMMARY:
Bacteria is occasionally present in the shoulder during shoulder arthroplasty surgery and is hypothesized to increase the risk of failure of the prosthesis. Surgiphor (sterile Povidone-Iodine) wound irrigation, is a solution used in orthopaedic surgery and other surgical fields to kill bacteria intraoperatively. The Iodine dissociates from complex and has antimicrobial properties, causing cell death of bacteria, fungi, and viruses through interactions with proteins, nucleotides, and fatty acids in the cytoplasm and cytoplasmic membrane.

This study examines the use of Povidone-Iodine during primary shoulder arthroplasty.

DETAILED DESCRIPTION:
The purpose of this study is to determine the rate of reduction of positive cultures collected before and after wound irrigation with either Surgiphor or sterile normal saline during primary total shoulder arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Adults age >18 years
* Participants undergoing elective primary total shoulder arthroplasty
* Participants willing to provide written consent

Exclusion Criteria:

* History of prior surgery to the operative shoulder
* Known allergy to povidone iodine, iodine or shellfish
* active clinical infection
* participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Reduction or elimination of bacteria | 90 days
  To determine the rate of reduction of positive cultures collected before and after wound irrigation with either Surgiphor or sterile normal saline during primary total shoulder arthroplasty participants will be followed to watch for clinical signs of infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No